CLINICAL TRIAL: NCT02117219
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of MEDI4736 as Monotherapy or in Combination With Tremelimumab With or Without Azacitidine in Subjects With Myelodysplastic Syndrome After Treatment With Hypomethylating Agents
Brief Title: Phase 1 Study to Evaluate MEDI4736 in Subjects With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00007
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — durvalumab; Azacitidine; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI4736 Evaluate MEDI4736 in MDS (Experimental): Evaluate MEDI4736 monotherapy and MEDI4736 in combination with azacitidine after monotherapy progression in MDS
  Interventions: Biological: MEDI4736 Evaluate MEDI4736 in MDS; Drug: VIDAZA
- MEDI4736 + tremelimumab (Experimental): Evaluate MEDI4736 in combination with tremelimumab
  Interventions: Biological: tremelimumab
- MEDI4736 + tremelimumab + azacitidine (Experimental): Evaluate MEDI4736 in combination with tremelimumab and azacitidine
  Interventions: Drug: VIDAZA; Biological: tremelimumab

INTERVENTIONS:
Biological: MEDI4736 Evaluate MEDI4736 in MDS — MEDI4736 will be administered by IV infusion
  Other Names: durvalumab
  Arms: MEDI4736 Evaluate MEDI4736 in MDS
Drug: VIDAZA — VIDAZA will be administered subcutaneously as described on the package insert VIDAZA will be administered in combination with MEDI4736 upon progression from MEDI4736 monotherapy
  Other Names: azacitidine
  Arms: MEDI4736 + tremelimumab + azacitidine; MEDI4736 Evaluate MEDI4736 in MDS
Biological: tremelimumab — tremelimumab will be administered by IV infusion
  Arms: MEDI4736 + tremelimumab; MEDI4736 + tremelimumab + azacitidine

SUMMARY:
This is a multicenter, open-label, Phase 1 study to assess the safety and antitumor activity of MEDI4736 as Monotherapy or in Combination with Tremelimumab with or without Azacitidine in Subjects with myelodysplastic syndrome after treatment with hypomethylating agents

DETAILED DESCRIPTION:
A dose-escalation and dose-expansion study of MEDI4736 (a monoclonal antibody that targets programmed cell death-1 ligand 1 [PD-L1]) to evaluate the safety, tolerability, PK, IM, and antitumor activity of MEDI4736 as monotherapy or in combination with Tremelimumab with or without Azacitidine in adult patients with myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

Adult male or female subjects with pathologically confirmed MDS who failed to respond, relapsed after an initial response, or were unable to tolerate hypomethylating agents, ECOG performance status of 0 - 2, and adequate organ and marrow function.

Exclusion Criteria:

Concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment, prior MAb against CTLA-4, PD-1, or PD-L1, alllogenic or haploidentical transplant, current immunosuppressive medication or autoimmune or inflammatory disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Subject's safety where no more than one out of six subjects experience DLTs at a given dose | 180 days
  DLT (MEDI4736 monotherapy only) assessment will be done by reviewing adverse events (AEs), serious adverse events (SAEs), laboratory evaluations, vital signs, physical examinations, and electrocardiogram (ECG) results. For monotherapy or combo w/aza AEs, SAEs, lab evaluations, vital signs, physical exams, ECGs will be done.
Subject's safety overall (monotherapy and combination therapies) | 730 days
  Overall safety assessments will be done by reviewing adverse events (AEs, serious adverse events (SAEs), laboratory evaluations, vital signs, physical examinations and electrocardiogram (ECG) results.

SECONDARY OUTCOMES:
Clinical outcome in terms of response: duration of response | 2 years
  As defined by IWG 2006 MDS response criteria
Clinical outcome in terms of response: transfusion requirements | 2 years
  As defined by IWG 2006 MDS response criteria and incidence of transfusions.
Clinical outcome in terms of response: progression-free survival (PFS) | 2 years
  As defined by IWG 2006 MDS response criteria
Clinical outcome in terms of response: survival (OS) | 2 years
  As defined by IWG 2006 MDS response criteria and collection of survival data
Pharmacokinetics: MEDI4736 and tremelimumab concentrations in serum: peak concentration | 1 year
  Peak concentration of MEDI4736 and tremelimumab in serum
Pharmacokinetics: MEDI4736 and tremelimumab concentrations in serum: area under the concentration-time curve | 1 year
  Analysis of area under the concentration-time curve
Pharmacokinetics: MEDI4736 and tremelimumab concentration in serum: clearance | 1 year
  Rate of MEDI4736 and tremelimumab clearance
Pharmacokinetics: MEDI4736 and tremelimumab concentration in serum: terminal half-life | 1 year
  MEDI4736 and tremelimumab concentration terminal half-life
Immunogenicity | 1 year
  Determine by number of subjects who develop ADA (anti-drug antibody).
Health-related quality of life (QOL): disease- and treatment-related symptoms (Part 1 only) | 2 years
  Analysis of reporting of disease- and treatment-related symptoms (Part 1 only)
Health-related quality of life (QOL): pain (Part 1 only) | 2 years
  Analysis of incidence of pain reporting (Part 1 only)
Health-related quality of life (QOL): health status (Part 1 only) | 2 years
  Analysis of reporting of health status. (Part 1 only)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (20):
- United States (15):
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Greenville, South Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Milwaukee, Wisconsin
- Research Site, Paris, France
- Research Site, Dresden, Germany
- United Kingdom (3):
  - Research Site, Brighton
  - Research Site, London
  - Research Site, Manchester